CLINICAL TRIAL: NCT06893952
Title: Technical Evaluation and Results of the Use of TREO® Modular Aortic Endografts for the Treatment of Abdominal Aortic Aneurysms
Acronym: RegisTREO
Status: Not yet recruiting | Type: Observational
Sponsor: Vascutek Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: RegisTREO _2024.01
Record Dates: First submitted 2025-02-17; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Aortic Aneurysm Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: TREO Endograft — Post Market collection data in use of TREO modular endografts

SUMMARY:
This study is a clinical investigation as part of the post-market clinical follow-up of the TREO® abdominal aortic graft in its initial use, French, observational, multicenter, non-randomized, single-arm. Information on patient's health and the implanted device will be collected over a period of 5 consecutive years. The data collected will be analyzed on the technical success and the absence of major events (death, stroke, myocardial infarction, visceral ischemia, paraplegia, respiratory failure, renal failure, intraoperative blood loss, thromboembolic event) and possible reinterventions related to the patient's operation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who has confirmed his/her non-opposition to the use of his/her data in the study.
2. Patient aged 45 years or older.
3. Patient with AAA with one of the following criteria:

   * Maximum diameter ≥50 mm for women and ≥55 mm for men
   * Rapid growth (≥5 mm in 6 months or ≥10 mm in 12 months)
   * Unruptured AAA with clinical symptoms of abdominal pain
4. Adequate anatomy for TREO® stent graft implantation, including:

   * Adequate iliac and femoral arteries for the modular system
   * Suprarenal angle less than 45 degrees
   * Infrarenal aortic neck greater than or equal to 10 mm in length with an angle less than 60° and an internal diameter of 17mm-32mm, or an infrarenal aortic neck greater than or equal to 15 mm in length with an angle between 60 and 75° and an internal diameter of 16mm-30mm
   * Distal iliac sealing distance ≥ 10 mm and an iliac diameter between 8-13 mm or a distal iliac sealing distance ≥ 15 mm and a diameter between 13-21 mm
5. Ability to follow the entire protocol from 1 to 60 months
6. Life expectancy greater than 2 years

Exclusion Criteria:

1. Patients refusing treatment and follow-up as part of the study
2. Infected or ruptured aneurysm
3. Associated aortic lesion (thoracic or thoracoabdominal aneurysm) requiring management
4. Renal failure defined by creatinine > 2.5 mg/dL or patient in pre-dialysis status and impossibility of intervention with use of CO2 injection
5. New York Heart Association (NYHA) class IV
6. Aneurysmal, dissected distal implantation zone, or including calcifications and/or significant thrombus that could compromise sealing
7. Tortuous iliac and/or femoral access and/or including calcified stenosis
8. Systemic infection that could increase the risk of infection of the endoprosthesis
9. Pathology of the supporting tissues such as collagenosis (Marfan or Ehler-Danlos, etc.)
10. Known drug use
11. Known sensitivity or allergy to the materials to be implanted
12. Patients contraindicated for antiplatelet treatment
13. Patients with an uncontrolled hematological disorder or heparin-induced thrombocytopenia
14. Patients who are pregnant or planning to become pregnant
15. Patients considered hemodynamically unstable or requiring emergency treatment
16. Patients with severe arterial disease leading to a negative "outflow" that may degrade the permeability of implanted stents
17. Scheduled hybrid aortic technique (surgical and endovascular)
18. Patients with complex iliac access outside the manufacturer's indications and recommendations that may lead to procedural failure

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with:
  * an asymptomatic infrarenal abdominal aortic aneurysm with a largest diameter greater than 5.5 cm in men and 5 cm in women or if the diameter increases by 1 cm in 1 year (for an aneurysm with a diameter greater than 4 cm).
  * a symptomatic infrarenal abdominal aortic aneurysm, regardless of the size.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcomes of this study are the rate of a composite measure of technical and clinical success at 1 and 12 months to assess efficacy, and the rate of a composite measure of free from major adverse events at 1 month to assess safety. | 12 months
  Definition of the composite of technical success:
  * Successful access to the arterial system using remote arterial exposure, percutaneous technique, surgical access, or open surgical conduits.
  * Successful delivery and deployment of all components of the modular stent graft.
  * Absence of type I or type III endoleaks at the end of angiography that extend beyond 30 days confirmed by imaging*.
  * Patency of all components of the modular stent graft.
  Definition of the composite of clinical success :
  * Technical success
  * No death during the initial procedure, related to the procedure or from aortic-related causes during the initial hospitalization
  * No type I and III endoleaks, at 1 and 12 months
  * No early migration (> 10 mm), at 1 and 12 months
  * No increase in maximum sac diameter of more than 5 mm between 1 and 12 months
  * No aneurysm rupture, at 1 and 12 months
  * No surgical conversion related to aneurysm treatment, at 1 and 12 months

IPD SHARING:
Plan to Share IPD: No